CLINICAL TRIAL: NCT04102137
Title: Antibody Persistence at 3 Years After a Single Dose Vaccination of Acellular Pertussis Vaccines Containing Genetically-detoxified Pertussis Toxin
Brief Title: 3-year Follow-up After a Single Dose Acellular Pertussis Vaccination
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Other Study IDs: TDA202 3 year follow-up
Record Dates: First submitted 2019-09-22; First posted 2019-09-25 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Pertussis
Keywords: TDA202; acellular pertussis vaccine; antibody persistence at 3 years after vaccination; Pertagen; Boostagen; aP vaccine
MeSH Terms: conditions — Whooping Cough | interventions — adacel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Approximately 5 mL whole blood will be processed for serum preparation. Sera obtained will be aliquoted into storage tubes and stored ≤ -60 degree Celsius and shipped to Bionet Human Serology Laboratory. The collected sera will be used for immunogenicity assessment for antibody persistence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3: Antibody persistence at 3 years after a single dose vaccination of acellular pertussis vaccines
  Interventions: Biological: Pertagen (aP BioNet); Biological: Boostagen (TDaP BioNet); Biological: Adacel

INTERVENTIONS:
Biological: Pertagen (aP BioNet) — Pertagen (aP BioNet) was produced with a recombinant B pertussis strain that was genetically inactivated by the introduction of mutations (Arg9Lys and Glu129Gly) in the ptx operon of the S1 gene. Each 0.5 mL dose of Pertagen (aP BioNet) contained 5 µg PTgen, 5 µg FHA, and 0.3 mg as aluminium cation.
  The study vaccine will be presented in a single-dose prefilled syringe. Each subject will be received one intramuscular injection in the non-dominant deltoid region.
Biological: Boostagen (TDaP BioNet) — Boostagen (TDaP BioNet) was produced with a recombinant B pertussis strain that was genetically inactivated by the introduction of mutations (Arg9Lys and Glu129Gly) in the ptx operon of the S1 gene. Each 0.5 mL dose of Boostagen (TDaP BioNet) contained 5 µg PTgen, 5 µg FHA, and 0.3 mg as aluminium cation. TDaP dose additional contained at least 7.5 Lf tetanus toxoid and at least 2.0 Lf diphtheria toxoid.
  The study vaccine will be presented in a single-dose prefilled syringe. Each subject will be received one intramuscular injection in the non-dominant deltoid region.
Biological: Adacel — Comparator vaccine, Adacel (Sanofi-Pasteur, North York, ON, Canada) was produced chemically inactivated pertussis toxin. Each 0.5 mL dose of Adacel (as comparator vaccine) contained 2.5 µg PTchem, 5 µg FHA, 3 µg pertactin, 5 µg fimbriae types 2 and 3, 5.0 Lf tetanus toxoid, 2.0 Lf diphtheria toxoid and 0.33 mg as aluminium cation.
  The study vaccine will be presented in a single-dose prefilled syringe. Each subject will be received one intramuscular injection in the non-dominant deltoid region.

SUMMARY:
In July 2015-November 2016, a phase II/III randomized, observer-blind,controlled study of two acellular Pertussis vaccines (aP standalone and TdaP combined vaccined) manufactured by BioNet-Asia Co., Ltd. (Bionet) and chemically-detoxified Adacel Tdap vaccine was conducted in Bangkok, Thailand in healthy subjects aged 12-17 years (Protocol No. TDA202; http://clinicaltrials.in.th;Study ID:TCTR20150703002). A total of 450 subjects were enrolled into the study at 2 study sites (Site No.1:Faculty of Medicine Siriraj Hospital; Site No.2:Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University) with equal number of 225 subjects enrolled at each study site. During the study, the subjects had been randomized in a 1:1:1 ratio to received intramuscularly a booster dose (0.5 mL) of the study vaccines.

This is further follow-up from TDA202 clinical trial, which was completed on 29 November 2016. Target population for this study is the group of subjects who had received one dose of one of the three study vaccines in the TDA202 trial at site VTC and who had completed the study follow-up at 1-year after vaccination (223 subjects).

In this current study, the long-term persistence of pertussis antibodies induced by a booster dose of recombinant acellular Pertussis based vaccines (Pertagen and Boostagen) manufactured by Bionet will be evaluated and compared to the conventional chemically-detoxified Tdap vaccine (Adacel) at 3 years after previously immunized in the TDA202 study.

DETAILED DESCRIPTION:
The study population will included all subjects who participated in the TDA202 study at the Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University, Bangkok.

The subjects who had received a single dose of one of the 3 study vaccines and completed 1-year follow-up visit at Day 336±28 during the TDA202 study will be called in for consent process at 3 years after vaccination based on Vaccination Date in TDA202 study within ±1 month window period. Subjects aged ≥ 18 years who have signed the written informed consent form or subjects aged < 18 years who have signed the assent form with their parent/legal guardian's given written informed consent will be screened for general health status and those who fulfill all inclusion and exclusion criteria will be enrolled into the study.

Once enrolled, blood sample (approximately 5 mL) will be taken from all subjects. After blood collection, vaccination with a licensed influenza vaccine will be offered to all subjects.Blood samples will be processed for serum separation and shipped to Bionet Human Serology Laboratory where immunogenicity testing (ELISA antibodies against tetanus (TT), diphtheria(DT), Pertussis Toxin (PT) and Filamentous hemagglutinin (FHA) and PT neutralizing antibody by Chinese Hamster Ovary (CHO cell assay) will be performed . ELISA testing to detect antibodies against tetanus, diphtheria, and pertussis antigens (PT and FHA) will be performed for all enrolled subjects while CHO cell assay to detect PT neutralizing antibody will be performed only in the same subset of 75 subjects (25 subjects in each vaccine group) who had been selected for PT neutralizing antibody assessment in the previous TDA202 study.

The knowledge from this long-term 3-year antibody persistence study will provide supportive data to identify the best alternative acellular pertussis vaccines to conventional chemically-detoxified vaccines for controlling the resurgence of pertussis disease.

Data management and statistical analysis will be performed by Center of Excellence for Biomedical and Public Health Informatics (BIOPHICS), Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Having participated in TDA202 study, received a single dose of one of the 3 study vaccines, and completed 1 year follow-up visit.
2. Written informed consent is obtained for subjects aged ≥18 years, or written assent and written informed consent are obtained from subjects aged <18 years and from their parent/legal guardian, respectively, prior to study entry.
3. Capable to comply with study procedures and willing to provide with a blood sample.

Exclusion Criteria:

No exclusion criteria for this study. Subjects will be eligible for participation if all inclusion criteria are met.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population for this study is the group of subjects who had received one dose of acellular pertussis based vaccine in TDA202 trial at Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University and who had completed the study follow-up at 1 year after vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Comparison of anti-PT GMTs (IU/mL) between baseline and 3 years after vaccination | 3 years after vaccination ± 1 month
  Assessed by ELISA in all evaluable subjects by vaccine groups
Comparison of anti-FHA GMTs (IU/mL) between baseline and 3 years after vaccination | 3 years after vaccination ± 1 month
  Assessed by ELISA in all evaluable subjects by vaccine groups
Comparison of anti-Tetanus GMTs (IU/mL) between Day 336 and 3 years after vaccination | 3 years after vaccination ± 1 month
  Assessed by ELISA in all evaluable subjects by vaccine groups
Comparison of anti-Diphtheria GMTs (IU/mL) between Day 336 and 3 years after vaccination | 3 years after vaccination ± 1 month
  Assessed by ELISA in all evaluable subjects by vaccine groups
Seroconversion rates of subjects with anti-PT antibody titers at 3 years after vaccination compared to baseline in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  Booster response:
  * In initially seronegative subjects (baseline titer < 5 IU/mL), post-vaccination antibody concentrations ≥ 20 IU/mL;
  * In initially seropositive subjects with baseline titer ≥ 5 IU/mL and < 20 IU/mL, an increase of at least 4 times (≥ 4-fold) the baseline titer;
  * In initially seropositive subjects with baseline titer ≥ 20 IU/mL, an increase of at least 2 times (≥ 2-fold) the baseline titer
Seroconversion rates of subjects with anti-FHA antibody titers at 3 years after vaccination compared to baseline in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  Booster response:
  * In initially seronegative subjects (baseline titer < 5 IU/mL), post-vaccination antibody concentrations ≥ 20 IU/mL;
  * In initially seropositive subjects with baseline titer ≥ 5 IU/mL and < 20 IU/mL, an increase of at least 4 times (≥ 4-fold) the baseline titer;
  * In initially seropositive subjects with baseline titer ≥ 20 IU/mL, an increase of at least 2 times (≥ 2-fold) the baseline titer
Seroconversion rates of subjects with ≥ 2-fold increase in anti-PT antibody titers at 3 years after vaccination compared to baseline, Day 336 and 2 years after vaccination in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  by ELISA in all evaluable groups
Seroconversion rates of subjects with ≥ 2-fold increase in anti-FHA antibody titers at 3 years after vaccination compared to baseline, Day 336 and 2 years after vaccination in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  by ELISA in all evaluable groups
Seroconversion rates of subjects with ≥ 4-fold increase in anti-PT antibody titers at 3 years after vaccination compared to baseline, Day 336 and 2 years after vaccination in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  by ELISA in all evaluable groups
Seroconversion rates of subjects with ≥ 4-fold increase in anti-FHA antibody titers at 3 years after vaccination compared to baseline, Day 336 and 2 years after vaccination in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  by ELISA in all evaluable groups
Seroconversion rates of subjects with > 0.1 IU/mL of anti-Tetanus at baseline and 3 years after vaccination compared to baseline in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  Assessed by ELISA
Seroconversion rates of subjects with > 0.1 IU/mL of anti-Diphtheria at baseline and 3 years after vaccination compared to baseline in all evaluable subjects by vaccine groups | 3 years after vaccination ± 1 month
  Assessed by ELISA
Comparison of PT neutralizing GMTs (IU/mL) between baseline and 3 year after vaccination | 3 years after vaccination ± 1 month
  PT neutralizing antibody assessed by Chinese Hamster Ovary (CHO) in subset of each vaccine group
Seroconversion rates of PT neutralizing antibody increase ≥ 4-fold at 3 years after vaccination compared to baseline, Day 336 and 2 years after vaccination | 3 years after vaccination ± 1 month
  PT neutralizing antibody assessed by Chinese Hamster Ovary (CHO) in subset of each vaccine group

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, Principal Investigator — VTC, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mhahidol University, 420/6 Ratchawithi Road, Ratchathewi,, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pitisuttithum P, Chokephaibulkit K, Sirivichayakul C, Sricharoenchai S, Dhitavat J, Pitisuthitham A, Phongsamart W, Boonnak K, Lapphra K, Sabmee Y, Wittawatmongkol O, Chauhan M, Wijagkanalan W, Hommalai G, Fortuna L, Chinwangso P, Poredi IK, van den Biggelaar AHJ, Pham HT, Viviani S. Antibody persistence after vaccination of adolescents with monovalent and combined acellular pertussis vaccines containing genetically inactivated pertussis toxin: a phase 2/3 randomised, controlled, non-inferiority trial. Lancet Infect Dis. 2018 Nov;18(11):1260-1268. doi: 10.1016/S1473-3099(18)30375-X. Epub 2018 Sep 25. PMID 30266329